CLINICAL TRIAL: NCT05614674
Title: The Examination of Relationship Between Self-Efficacy and Sensorial, Perceptual and Motor Skills in People With Chronic Low Back Pain A Cross-Sectional Study
Brief Title: The Examination of Relationship Between Self-Efficacy in People With Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Burak Kara, Physiotherapist, Suleyman Demirel University
Other Study IDs: 72867572-050.01.04-379338
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Self Efficacy
Keywords: Back Pain; Propioception; Depression; Pain Catastrophizing; Flexibility; Balance
MeSH Terms: conditions — Back Pain; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: People who don't suffer from low back pain
- People with low back pain: People who are suffering from low back pain. The pain level has to be at least 3 out of 10 according to Visual Analog Scale (VAS) to be in this group.

SUMMARY:
Self-efficacy is defined as a person's confidence or belief that one can achieve a certain behavioral or cognitive state. Self-efficacy is one of the most important assesment parameters in the self-management model. It is accepted that patients with chronic low back pain with high self-efficacy have a better prognosis than those with low self-efficacy. Due to the complex nature of pain; The relationship between psychological and physical parameters such as pain catastrophy, disability level, depression, physical performance, self-efficacy, pain intensity and fear avoidance arouses curiosity. The aim of this cross-sectional study is to examine the relationship between the level of self-efficacy and sensory, perceptual and motor skills in people with chronic low back pain.

ELIGIBILITY:
Inclusion Criterias For Healthy Group:

* Being minimum 30 maximum 65 years old
* To be literate
* Accepting to take part in the study

Inclusion Criterias For Partipicians with Low Back Pain Group:

* Being minimum 30 maximum 65 years old
* Minimum 3 score from Visual Analog Scale (VAS)
* Having low back pain for at least 3 months of time
* To be literate
* Accepting to take part in the study

Exclusion Criteria:

* Any kind of surgery in low back area
* Surgery story in lower extremities
* Acute low back pain
* Having a neurological disorder
* Having a rheumatological disease which may cause to low back pain
* Having a herniated disc that presses on the sacral nerves
* Being pregnant

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study group will consist of 30-65 years old people who will be agreed to take part in the study. There will be two groups. 1 of them is healthy group and the other is for people with low back pain. The partipicians will be literate enough to answer the questions in scales and questionnares by themselves
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline
Proprioception Measurement with G-Pro Phone App | Baseline
Beck Depression Inventory (BDI) | Baseline
Pain Catastrophizing Scale (PCS) | Baseline
Sit and Reach Test (SRT) | Baseline
Multidirectional Reach Test | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Burak Kara, Bachelor, Principal Investigator — Suleyman Demirel University